CLINICAL TRIAL: NCT06098638
Title: Effect of Aerobic and Resisted Exercise on Lipid Profile and Quality of Life in Overweight Breastfeeding Women: A Randomized Clinical Trial
Brief Title: Effect of Aerobic and Resisted Exercise on Lipid Profile and Quality of Life in Overweight Breastfeeding Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Gamal Mohamed Ali, physical therapist at Abo Kabir general hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No:P.T.REC/012/004227
Record Dates: First submitted 2023-10-14; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Postpartum Weight Retention
Keywords: exercise; breastfeeding; Overweight; lipid; life quality
MeSH Terms: conditions — Gestational Weight Gain; Motor Activity; Breast Feeding; Overweight

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: double (participant, outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Group (A) included 27 overweight breastfeeding woman who received nutritional recommendation and faradic current stimulation on the abdominal surface for 12 weeks, while group
  Interventions: Other: Nutritional recommendation and Faradic stimulation program
- exercise group (Experimental): Group (B) 27 overweight breastfeeding women, who received the same nutritional recommendation and faradic current stimulation on the abdominal surface plus exercise training (aerobic + resisted) for 12 weeks.
  Interventions: Other: Nutritional recommendation and Faradic stimulation program; Other: aerobic and resisted exercise for 12 weeks

INTERVENTIONS:
Other: Nutritional recommendation and Faradic stimulation program — proper maternal nutrition and fluid intake during breast-feeding per day for 12 weeks and2 sessions per week, each session 20 minutes, for 12 weeks. Frequency of 65 Hz, and width pulse 300 ms, with contraction time 10 sec and relaxation time 10 sec
Other: aerobic and resisted exercise for 12 weeks — Each woman in group (B) participated in a moderate exercise program (aerobic+resistive), 3 days/week, for 12 weeks. The session began with 15 minutes of aerobic exercise on a bicycle ergometer, at 60% of heart rate reserve (HRR), with HRR estimated (220-age-resting heart rate). Then, the participant was performed 15 minutes of resistive exercise (two sets of 8-12 repetitions at 75% of one repetition maximum (1-RM) for basic core exercises in the form of hip lifts, knee extension and flexion, crunches, shoulder flexion and extension, elbow flexion and extension with resistance
  Arms: exercise group

SUMMARY:
the aim of the study was to investigate the effect of aerobic and resisted exercise program on lipid profile and quality of life in overweight breastfeeding women.

DETAILED DESCRIPTION:
Although previous studies reported that exercise training during the postpartum period could improve the lipid profile and quality of life in overweight women and reduce the postpartum fatigue . None of them had investigated the effect of aerobic and resisted exercises on lipid profile and quality of life in overweight breastfeeding women.this trial will include 2 groups:

Group (A): was consist of 27 overweight breastfeeding women, who received nutritional recommendation and faradic current stimulation for 20 min on abdominal surface 2 times per week for 12 weeks.

Group (B): was consist of 27 overweight breastfeeding women, who received the same nutritional recommendation and faradic current stimulation for 20 min on abdominal surface 2 times per week plus exercise training (aerobic + resisted) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. All of women were sedentary, non-smoking, breastfeeding women at their 3rd to 6th months postpartum
2. they had delivered a single, healthy, mature fetus with no complications through normal vaginal delivery.
3. Their age was ranged from 20 to 30 years old.
4. Their parity number was one or two.
5. They were overweight (body mass index (BMI) was ranged from 25 to 30 kg/m²).

Exclusion Criteria:

1. Having chronic disorders, heart disease, respiratory infections, diabetes mellitus, pelvic abnormalities, hormonal abnormalities, psychological problems, menstrual disorders or anemia of other pathological origins.
2. Receiving any type of physical exercise or sport.
3. Following a specific diet program.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female (overweight breast feeding)
Enrollment: 54 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
measurement of lipid parameter level of High-density lipoprotein (HDL) mg/dL | 12 weeks
  It was used to measure the lipid profile parameters (High-density lipoprotein (HDL)- level in for each woman in the both groups (A & B) at pre-treatment and post-treatment.
measurement of Low-density lipoprotein (LDL) mg/dL | 12 weeks
  It was used to measure the lipid profile parameters Low-density lipoprotein (LDL) level for each woman in the both groups (A & B) at pre-treatment and post-treatment.
measurement of Triglycerides (TG) mg/dL | 12 weeks
  t was used to measure the lipid profile parameters Triglycerides (TG) level for each woman in the both groups (A & B) at pre-treatment and post-treatment.

SECONDARY OUTCOMES:
calculation of score of Short Form 36 Health Survey Questionnaire (SF-36) (Arabic version): | 12 weeks
  It was assessed using the SF-36 (Arabic version) questionnaire in both groups (A & B) before and after treatment, which consists of 36 questions. Answers were awarded a score in a five-point scale (0-4).Scores for each of the dimensions range from 0 (worst level of functioning) to 4 (best level of functioning)

OTHER OUTCOMES:
body mass index (BMI) kg/m² | 12 weeks
  The height and weight were determined for each woman in the both groups (A & B) to calculate her (BMI = (weight in kg)/(height in m^2 ) ) at pre-treatment and post-treatment
waist to hip ratio (W/H ratio) | 12 weeks
  The waist and hip circumferences were taken for each woman in both groups (A & B) before and after treatment course for calculating waist and hip ratio (W/H ratio) by dividing waist circumference (WC) on the hip circumference (HC).

CONTACTS AND LOCATIONS:
Overall Officials: marwa G anany, Principal Investigator — Cairo University
Locations (1):
- Marwa Gamal Mohamed Ali Anany, Abū Kabīr, Abu Kabir, Egypt

IPD SHARING:
Plan to Share IPD: No